CLINICAL TRIAL: NCT05634629
Title: Anterior Lamellar Recession vs Bilamellar Tarsal Rotation in Upper Lid Cicatricial Trichiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab tharwat, Principal Investigator, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cicatricial trichiasi
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Cicatricial Trichiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Lamellar Recession (Active Comparator)
  Interventions: Procedure: Anterior Lamellar Recession
- Bilamellar Tarsal Rotation (Active Comparator)
  Interventions: Procedure: Bilamellar Tarsal Rotation

INTERVENTIONS:
Procedure: Anterior Lamellar Recession — ALR is a common surgical treatment that splits the skin and orbicularis oculi muscle from the tarsus and conjunctiva to recede the anterior lamella and expose the tarsus. Interlamellar separation can be accomplished via a grey line technique, an eyelid crease approach, or a combination of the two
  Arms: Anterior Lamellar Recession
Procedure: Bilamellar Tarsal Rotation — the full-thickness transverse blepharotomy combined with everting sutures to rotate the inferior portion of the upper lid outwards and this procedure has a low recurrence risk
  Arms: Bilamellar Tarsal Rotation

SUMMARY:
in recent years there has been a significant shift from this destructive procedure to a reconstructive procedure such as Anterior Lamellar Recession (ALR) and Bilamellar Tarsal Rotation (BLTR).

ELIGIBILITY:
Inclusion Criteria:

* patients with upper lid cicatricial trichiasis that requires surgical intervention

Exclusion Criteria:

* Refusal of the patients.
* Associated entropion., 3) Severe ocular surface disease.
* Previous eyelid surgery.
* Associated lid laxity.
* Lack of adequate follow-up

Ages: 48 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
lid correction | at 1 month post operative
  Its a subjective outcome that will be collected through an interview after the surgery. it consists of 3 sub domaines which include (adequate correction, undercorrection, and over corrections)
lid correction | 3 months postoperative
  Its a subjective outcome that will be collected through an interview after the surgery. it consists of 3 sub domaines which include (adequate correction, undercorrection, and over corrections)
lid correction | 6 months postoperative
  Its a subjective outcome that will be collected through an interview after the surgery. it consists of 3 sub domaines which include (adequate correction, undercorrection, and over corrections)
Cosmetic Satisfaction | at 1 months post operative
  Its a subjective outcome that will be collected through an interview after the surgery.
Cosmetic Satisfaction | at 3 months post operative
  Its a subjective outcome that will be collected through an interview after the surgery.
Cosmetic Satisfaction | at 6 months post operative
  Its a subjective outcome that will be collected through an interview after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided